CLINICAL TRIAL: NCT05039827
Title: Comparison Of Mobilization With Movement And Soft Tissue Mobilization On Pain Severity , Hand Grip Strength And Functional Activity Tennis Elbow Patients.
Brief Title: Mobilition With Movement and Soft Tissue Mobiiztion in Tennis Elbow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/21/0420
Record Dates: First submitted 2021-09-01; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Tennis Elbow
MeSH Terms: conditions — Tennis Elbow | interventions — Movement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MWM GROUP (Experimental): Mobilization with movement with wrist extension
  Interventions: Other: Mobilization with movement
- SOFT TISSUE MOBILIZATION GROUP (Active Comparator): Parallel and perpendicular soft tissue massage at common extensor origin
  Interventions: Other: Soft Tissue Mobilization

INTERVENTIONS:
Other: Mobilization with movement — Heating fermentation was done for 10 minutes as baseline treatment. MWM with wrist extension was given for alternative days in a week as per 3 sessions per week for 4 weeks.
  Arms: MWM GROUP
Other: Soft Tissue Mobilization — Heating fermentation was done for 10 minutes as baseline treatment. Parallel and longitudinal massage was given for alternative days in a week as per 3 sessions per week for 4 weeks
  Arms: SOFT TISSUE MOBILIZATION GROUP

SUMMARY:
Lateral epicondylitis or tennis elbow is one of the most common lesions of the arm. This injury is a major challenge, as it is difficult to treat, prone to recurrence and may last for several weeks or months, with an average duration of a typical episode which has been reported to be between six months to two years. This is an RCT study. Subjects who fulfilled inclusion criteria will be taken for the study. Before conducting the actual method for subjects, lateral epicondylitis evaluation is done. First day before treatment, pain evaluation were done by using Numeric Pain Rating Scale. Muscle power was assessed by MMT (Manual Muscle Testing) and the function level are tested by Patient-Related Tennis Elbow Evaluation (PRTEE) questionnaire and asked to mark the results. Subjects will be divided into 2 groups randomly by lottery method. Each group consists of 15 patients. Group A will be given MWM; Group B will be given soft tissue mobilization. Both groups will be given with the above said methods for alternative days in a week as per 3 sessions per week for 4 weeks. At the end of program subjects will be reassessed by recording muscle strength, pain intensity and functional level. Finally pre and post recordings will be compared and analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Tennis players.
* Age group between 15-30 years.
* Positive specific tests.(cozen and mills test)
* Subjects having lateral epicondylitis pain for at least 4 weeks, muscle power for wrist muscle should be increase with activity against resistance, average pain level of 3-cm or more on a 10-cm Numerical pain rating scale

Exclusion Criteria:

* Any neurological disorder.
* Other elbow deformity or joint pathology. fracture of upper limb

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4 Week
  The Numeric Pain Rating Scale (NPRS) (an outcome measure) that is a unidimensional measure of pain intensity in adults.The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Grip Strength | 4 week
  Manual muscle testing as used to test grip strength. It involves testing key muscles from the upper and lower extremities against the examiner's resistance and grading the patient's strength on a 0 to 5 scale accordingly[1]:
  Flicker of movement Through full range actively with gravity counterbalanced Through full range actively against gravity Through full range actively against some resistance Through full range actively against strong resistance
Functional activity | 4 weeks
  Patient Related Tennis Elbow Evaluation (PRTEE) was used.The PrTEEQ is a 15-item questionnaire, it's designed to measure forearm pain and disability in patients with lateral epicondylitis. The patients have to rate their levels of tennis elbow pain and disability from 0 to 10, and consists of 2 subscales. There is the pain subscale (0 = no pain, 10 = worst imaginable) en the function subscale (0 = no difficulty, 10 = unable to do)

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Shafique, tDPT, Principal Investigator — Riphah International University
Locations (1):
- Hidayat Gillani Orthopedic Complex Sahiwal, Sahiwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bisset L, Paungmali A, Vicenzino B, Beller E. A systematic review and meta-analysis of clinical trials on physical interventions for lateral epicondylalgia. Br J Sports Med. 2005 Jul;39(7):411-22; discussion 411-22. doi: 10.1136/bjsm.2004.016170. PMID 15976161
- [Background] Castillo-Lozano R, Casuso-Holgado MJ. Incidence of musculoskeletal sport injuries in a sample of male and female recreational paddle-tennis players. J Sports Med Phys Fitness. 2017 Jun;57(6):816-821. doi: 10.23736/S0022-4707.16.06240-X. Epub 2016 Feb 12. PMID 26954572
- [Background] Lucado AM, Dale RB, Vincent J, Day JM. Do joint mobilizations assist in the recovery of lateral elbow tendinopathy? A systematic review and meta-analysis. J Hand Ther. 2019 Apr-Jun;32(2):262-276.e1. doi: 10.1016/j.jht.2018.01.010. Epub 2018 Apr 26. PMID 29705077
- [Background] Ahmed A, Ibrar M, Arsh A, Wali S, Hayat S, Abass S. Comparing the effectiveness of Mulligan mobilization versus Cyriax approach in the management of patients with subacute lateral epicondylitis. J Pak Med Assoc. 2021 Jan;71(1(A)):12-15. doi: 10.47391/JPMA.186. PMID 33484510
- [Background] Coombes BK, Connelly L, Bisset L, Vicenzino B. Economic evaluation favours physiotherapy but not corticosteroid injection as a first-line intervention for chronic lateral epicondylalgia: evidence from a randomised clinical trial. Br J Sports Med. 2016 Nov;50(22):1400-1405. doi: 10.1136/bjsports-2015-094729. Epub 2015 Jun 2. PMID 26036675